CLINICAL TRIAL: NCT03008408
Title: A Phase II, Randomized Two-Arm Study of Everolimus and Letrozole, +/- Ribociclib (LEE011) in Patients With Advanced or Recurrent Endometrial Carcinoma
Brief Title: A Phase II, Two-Arm Study of Everolimus and Letrozole, +/- Ribociclib (Lee011) in Patients With Advanced or Recurrent Endometrial Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0961; NCI-2018-01284 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0961 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-12-28; First posted 2017-01-02 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Recurrent Endometrial Carcinoma; Recurrent Endometrial Endometrioid Adenocarcinoma; Refractory Endometrial Carcinoma; Refractory Endometrial Endometrioid Adenocarcinoma; Stage III Uterine Corpus Cancer AJCC v8; Stage IIIA Uterine Corpus Cancer AJCC v8; Stage IIIB Uterine Corpus Cancer AJCC v8; Stage IIIC Uterine Corpus Cancer AJCC v8; Stage IIIC1 Uterine Corpus Cancer AJCC v8; Stage IIIC2 Uterine Corpus Cancer AJCC v8; Stage IV Uterine Corpus Cancer AJCC v8; Stage IVA Uterine Corpus Cancer AJCC v8; Stage IVB Uterine Corpus Cancer AJCC v8
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Everolimus; Letrozole; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (ribociclib, everolimus, letrozole) (Experimental): Patients receive ribociclib PO QD, everolimus PO QD, and letrozole PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Everolimus; Drug: Letrozole; Drug: Ribociclib
- Arm II (everolimus, letrozole) (Experimental): Patients receive everolimus PO QD and letrozole PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Everolimus; Drug: Letrozole

INTERVENTIONS:
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001; Votubia; Zortress
Drug: Letrozole — Given PO
  Other Names: CGS 20267; Femara
Drug: Ribociclib — Given PO
  Other Names: Kisqali; LEE-011; LEE011
  Arms: Arm I (ribociclib, everolimus, letrozole)

SUMMARY:
This phase II trial studies how well everolimus and letrozole with or without ribociclib work in treating participants with endometrial cancer that has spread to other areas of the body or has come back. Ribociclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs such as everolimus and letrozole have been shown to be effective at stopping tumor growth either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ribociclib, everolimus, and letrozole may work better than everolimus and letrozole in treating participants with endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the addition of ribociclib (LEE011) to everolimus and letrozole improves progression free survival in patients with advanced or recurrent endometrial carcinoma.

SECONDARY OBJECTIVES:

I. To determine clinical benefit and the median duration of progression-free survival (PFS) and overall survival (OS) in patients with advanced or recurrent endometrial carcinoma treated with ribociclib (LEE011), everolimus and letrozole versus everolimus and letrozole alone.

II. To determine the frequency and severity of toxicities associated with ribociclib (LEE011), everolimus (RAD001), and letrozole in this cohort of patients.

III. To determine the presence of a CTNNB1 mutation is associated with response to ribociclib (LEE011), everolimus (RAD001), and letrozole.

IV. To determine if liquid biopsies at baseline and 8 weeks correlate with presence of a tissue mutation or response to therapy.

EXPLORATORY OBJECTIVE:

I. To examine the pharmacokinetic and pharmacodynamic effects of ribociclib in patients with advanced or recurrent endometrial carcinoma.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive ribociclib orally (PO) once daily (QD), everolimus PO QD, and letrozole PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive everolimus PO QD and letrozole PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 30 days and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed the informed consent (ICF) prior to any screening procedures being performed and is able to comply with protocol requirements.
* Patients must have histologically-confirmed endometrial carcinoma (endometrioid and mixed endometrioid tumors, any grade).
* Patients must have advanced or recurrent disease that is refractory to curative treatment based on imaging or clinical exam.
* Patient must consent to allow for a baseline tumor biopsy. Tumor material from biopsies done before the screening period are acceptable if the biopsy was performed within 3 months prior to the planned treatment start and no other systemic cancer therapy was administered in the interim. If a biopsy is performed and the specimen is considered non-diagnostic, does not have enough tissue, or the biopsy is deemed infeasible to perform, this does not prevent the patient from proceeding with the treatment
* Patients must have had no more than two prior chemotherapeutic regimens for recurrent endometrial carcinoma. Chemotherapy administered in conjunction with primary radiation as a radio-sensitizer is not counted as a prior treatment for recurrent or advanced disease.
* Prior radiation therapy of any kind is allowed.
* Prior treatment with letrozole is allowed if the patient meets the washout period of 10 days.
* All patients must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 defined as at least one "target lesion" that can be accurately measured in at least one dimension (>= 10 mm longest dimension to be recorded; Lymph nodes must be >= 15 mm per short axis). Each lesion must be > 20 mm when measured by palpation or conventional imaging techniques (computed tomography [CT] or magnetic resonance imaging [MRI] - based on primary physician preference) or > 10 mm with spiral CT scan. Measurable lesions must be at least 2 times the slice thickness in millimeters. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented. Ascites and pleural effusions are not considered measurable disease. If the measurable disease is confined to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology.
* Patients must not be pregnant, breastfeeding or of child-bearing potential. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a total hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal for greater than 12 months (if patient is uncertain of amenorrhea for 12 months, a pregnancy test will be done to confirm pregnancy status). Patients in whom ovaries are present and were not previously menopausal at the time of hysterectomy, should have a serum estradiol < 10 pm/mL to confirm ovarian senescence.
* Patients must be off all other anti-tumor therapies (including immunologic agents) for at least four weeks prior to study registration. Patients on hormonal agents require a washout for 10 days.
* Gynecologic Oncology Group (GOG) performance status of 0 to 1.
* Absolute neutrophil count >= 1.5 x 10^9/L (at screening).
* Platelets >= 100 x 10^9/L (at screening).
* Hemoglobin >= 9.0 g/dL (at screening).
* International normalized ratio (INR) =< 1.5 (at screening).
* Serum creatinine =< 1.5 mg/dL or creatinine clearance >=50 mL/min (at screening).
* Estimated glomerular filtration rate (eGFR) >= 30mL/min/1.73m^2 (at screening) according to the Modification of Diet in Renal Disease (MDRD) formula.
* In the absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x upper limit of normal (ULN). If the patient has liver metastases, ALT and AST < 5 x ULN (at screening).
* Total bilirubin < ULN; or total bilirubin =< 3.0 x ULN or direct bilirubin =< 1.5 x ULN in patients with well-documented Gilbert's syndrome (at screening).
* Fasting serum cholesterol =< 240 mg/dL or =< 7.75 mmol/L and fasting triglycerides =< 2.5 x ULN (at screening).

  * NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* Patient with available standard 12-lead electrocardiography (ECG) with the following parameters at screening: a. Corrected QT interval by Fridericia's formula (QTcF) interval at screening < 450 msec (using Fridericia's correction). b. Resting heart rate 50-100 beats per minute (bpm).

Exclusion Criteria:

* Patients who have uterine sarcomas, carcinosarcomas, serous tumors (any component) or pure clear cell carcinomas.
* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, etc.)
* Patient has not recovered from all toxicities related to prior anticancer therapies to National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 grade =< 1 (exception to this criterion: patients with grade 1 taxane-induced neuropathy, any grade of alopecia, amenorrhea or other toxicities not considered a safety risk for the patient as per investigator's discretion are allowed to enter the study).
* Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered as major surgery).
* Participation in other studies involving investigational drug(s) within 30 days prior to randomization or within 5 half-lives of the investigational product (whichever is longer) or participation in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical, short duration (< 5 days) of systemic corticosteroids, eye drops, local injections, or inhaled corticosteroids are allowed.
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period. Close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, bacillus Calmette-guerin (BCG), yellow fever, varicella and TY21a typhoid vaccines.
* Patients with central nervous system (CNS) involvement unless they meet all of the following criteria:

  * At least 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment.
  * Clinically stable CNS tumor at the time of screening and not receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases.
* Patient has a concurrent malignancy or malignancy within 3 years prior to starting study drug, with the exception of adequately treated, basal or squamous cell carcinoma curatively resected cervical cancer in situ.
* Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, may cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.).
* Patient has a known history of human immunodeficiency virus (HIV) infection (testing not mandatory).
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormalities, including any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to screening.
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV).
  * Documented cardiomyopathy.
  * Left ventricular ejection fraction (LVEF) < 50% as determined by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO) at screening.
  * Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g. bifascicular block, Mobitz type II and third-degree AV block).
  * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

    * Risk factors for Torsades de Pointe (TdP) including uncorrected hypocalcemia, hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.
    * Concomitant use of medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued (within 5 half-lives or 7 days prior to starting study drug) or replaced by safe alternative medication.
    * Inability to determine the QT interval on screening (QTcF, using Fridericia's correction).
    * Systolic blood pressure (SBP) > 160 mmHg or < 90 mmHg at screening.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study medication (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection associated with malabsorption).
* Patient is currently receiving any of the following medications and cannot be discontinued 7 days prior to starting study drug:

  * Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pummelos, star-fruit, and Seville oranges.
  * That have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5.
  * Herbal preparations/medications, dietary supplements.
  * Hormone replacement therapy, topical estrogens (including any intra-vaginal preparations), megestrol acetate and selective estrogen-receptor modulators (e.g. raloxifene).
* Patient is currently receiving warfarin or other coumarin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed.
* Liver disease such as cirrhosis or severe hepatic impairment (patient with a Child-Pugh score B or C).

  * Note: A detailed assessment of hepatitis B/C medical history and risk factors must be done at screening for all patients. Hepatitis B virus (HBV) deoxyribonucleic acid (DNA) and hepatitis C virus (HCV) ribonucleic acid (RNA) polymerase chain reaction (PCR) testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection.
* Patients who have received prior treatment with an mTOR inhibitor (e.g., sirolimus, temsirolimus, everolimus).
* Patients with a known hypersensitivity to ribociclib or everolimus or to its excipients.
* History of noncompliance to medical regimens.
* Patients unwilling to or unable to comply with the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit rate (CBR) | At 8 weeks
  Per Response Evaluation Criteria in Solid Tumors version 1.1. This will be determined by combining the complete response rate, partial response rate, and stable disease rate. Response will be evaluated by repeat imaging (computed tomography or magnetic resonance imaging). Fisher's exact test will be used to compare patients with/without CTNNB1 mutation with respect to CBR.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela T Soliman, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org